CLINICAL TRIAL: NCT06835855
Title: Development of Attentional Biases for Affective Cues in Infants of Mothers With Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Binghamton University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00004999; R01MH132667 (NIH)
Record Dates: First submitted 2025-01-17; First posted 2025-02-19 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Depression - Major Depressive Disorder
Keywords: postpartum; infant; attention; psychophysiology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental protocol for all infants (Experimental)
  Interventions: Other: Passive Viewing Task; Other: Interaction Task

INTERVENTIONS:
Other: Passive Viewing Task — Infants will complete a computer-based task in which they view facial displays of emotion (angry, happy, sad, neutral) while an eye tracker records their gaze.
Other: Interaction Task — Mother and infants will also complete a standardized interaction task during which we assess infant gaze and psychophysiology. The task consists of three stages, each of which lasts three minutes. For the first stage (Free Play 1), infants sit in a highchair and mothers are asked to play with their baby as they normally would, without any toys or other objects. In the second stage (Sad), mothers are asked to think about times when they are sad or depressed and do not feel able to effectively play with their child. They are instructed to look at their child but speak in a monotone and minimize body movement or any physical contact with the infant. In the third stage (Free Play 2), mothers again interact with their infants normally for three minutes.

SUMMARY:
The goal of this study is to examine attentional biases for facial displays of emotion as a mechanism of risk in infants of mothers with postpartum major depression, and the potential role of infant arousal in the development of these attentional biases.

DETAILED DESCRIPTION:
As part of the study protocol, infants will complete a computer-based task in which they view facial displays of emotion (angry, happy, sad, neutral) while an eye tracker records their gaze. Mother and infants will also complete a standardized interaction task during which the investigators assess infant gaze and psychophysiology. The task consists of three stages, each of which lasts three minutes. For the first stage (Free Play 1), infants sit in a highchair and mothers are asked to play with their baby as they normally would, without any toys or other objects. In the second stage (Sad), mothers are asked to think about times when they are sad or depressed and do not feel able to effectively play with their child. Mothers are instructed to look at their child but speak in a monotone and minimize body movement or any physical contact with the infant. In the third stage (Free Play 2), mothers again interact with their infants normally for three minutes. These two tasks are consistent with the definition of a Basic Experimental Study in Humans (BESH).

ELIGIBILITY:
Inclusion Criteria:

* The high-risk group (n = 150) will consist of women with at least one episode of MDD since their baby's birth.
* To qualify for the low-risk group (n = 75), women cannot have a history of any depressive disorder or any current psychiatric diagnoses.
* Infants will be required to be singleton children born full-term (> 37 weeks) and normal weight (> 2,500 grams) with no birth complications or health problems to avoid medical complications contributing to infants' attention, reactivity, and regulation measures.
* The two groups will be matched on demographic factors (e.g., age, race/ethnicity, income).

Exclusion Criteria:

* Additional exclusion criteria are diagnoses of alcohol or substance use disorders currently or at any point during pregnancy, or lifetime history of bipolar or psychotic disorders.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Eye gaze during computer-based task | Baseline and 3-, 6-, 9-, and 12-month follow-up
  Used to determine percent of infant attention allocated to each emotional stimulus type (angry, happy, sad, neutral) during the computer-based task
Eye gaze during the interaction task | Baseline and 3-, 6-, 9-, and 12-month follow-up
  Used to assess the proportion of time during each phase of the interaction task that babies look at their mother (versus away from their mother)
Infant Heart Rate | Baseline and 3-, 6-, 9-, and 12-month follow-up
  During the interaction tasks, the investigators will record infant electrocardiography (ECG) to calculate heart rate (HR) using a MindWare Mobile system.
Infant Respiratory Sinus Arrhythmia | Baseline and 3-, 6-, 9-, and 12-month follow ups
  During the interaction tasks, the investigators will record infant electrocardiography (ECG) to calculate respiratory sinus arrhythmia (RSA) using a MindWare Mobile system. To calculate RSA, spectral power analyses will be performed with a fast Fourier transformation. RSA will be defined as power density in the .24-1.04 Hz frequency band and will be calculated for each 30 s epoch of each task.

SECONDARY OUTCOMES:
Infant social-emotional problems | Baseline and 3-, 6-, 9-, and 12-month follow-ups
  Infants' social-emotional problems will be assessed using mother reports on the Ages and Stages Questionnaire: Social-Emotional, Second Edition (ASQ:SE-2). Higher scores on the ASQ:SE-2 reflect greater social-emotional problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Binghamton University, Binghamton, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared via the NIMH Data Archive (NDA). All data will be de-identified prior to submission to the repository, but the information needed to generate a global unique identifier for the NDA will be collected for each subject.
Time Frame: All data will be deposited to NDA starting 12 months after the award begins and will be deposited every six months thereafter following the usual NDA data submission dates.
Access Criteria: Data will be findable for the research community through the NDA Collection that established when this application was funded. For all publications, an NDA study will be created. Each of those studies is assigned a digital object identifier (DOI). This data DOI will be referenced in the publication to allow the research community easy access to the exact data used in the publication.
URL: https://nda.nih.gov/edit_collection.html?id=5466